CLINICAL TRIAL: NCT06597448
Title: Public Health Nurse-Peer Co-Delivered Group Cognitive Behavioral Therapy for Postpartum Depression: A Randomized Controlled Trial
Brief Title: Public Health Nurse-Peer Co-Led Group Cognitive Behavioral Therapy for Postpartum Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Niagara Region Public Health (Other)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHN-Peer Co-Led CBT for PPD
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Depression
Keywords: Postpartum depression, PPD; Cognitive Behavioural Therapy; Public Health Nurse; Peer
MeSH Terms: conditions — Depression, Postpartum | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants who have met the eligibility requirements and signed the consent form are randomized and allocated in a 1:1 ratio to one of two groups: Intervention (those who participate in the 9-week CBT group along with treatment as usual) and Control (continue with treatment as usual alone). Control group participants receive a list of mental health resources. Both groups complete online questionnaires at 3 timepoints: enrollment (T1), 9 weeks later (T2-post intervention for those in the intervention group) and 6 months later (T3).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data analysts will be blinded. Data is deidentified and a study ID number is assigned. Research assistants following up with T2 and T3 questionnaires and phone interviews will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online CBT Group (Experimental): Participants randomized to the Intervention group will attend a 9-week online CBT group co-led by a Public Health Nurse and a Peer (individual who has recovered from PPD and received training to deliver the intervention) in addition to receiving usual care.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Postpartum Depression (PPD)
- Treatment as Usual (No Intervention): Participants randomized to the No Intervention group will continue to receive treatment as usual (standard postnatal care). A list of resources will be emailed.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Postpartum Depression (PPD) — Cognitive Behavioral Therapy (CBT) is a type of psychotherapy (talk therapy). The intervention consists of 9- 2hr sessions, the first half involves teaching and practice of CBT skills (cognitive restructuring, thinking errors, problem solving etc) followed by one hour of unstructured discussion around topics relevant to participants with Postpartum Depression (PPD) (sleep, supports, transitions, etc). Each group will be delivered by one randomly selected PHN and one randomly selected peer using our intervention manual.
  Arms: Online CBT Group

SUMMARY:
The purpose of this study is to determine the effectiveness of an online 9-week group Cognitive Behavioural Therapy (CBT; a type of talking therapy) intervention that is co-led by public health nurses (PHNs) and individuals who have previously recovered (i.e., lay peers) from postpartum depression (PPD) for treating PPD when delivered in addition to treatment as usual (TAU) compared to TAU alone. The study will also assess the impact of the intervention on common comorbidities (anxiety) and complications (parenting stress, mother-infant relationship, social support, and infant temperament) of PPD and whether it is cost-effective.

DETAILED DESCRIPTION:
The primary objective of the Randomized Controlled Trial (RCT) is to determine if a 9-week group Cognitive Behavioral Therapy (CBT) intervention delivered online and co-led by public health nurses (PHNs) and peers added to treatment as usual (TAU) can improve postpartum depression (PPD) more than TAU alone. Peers are individuals who have previously recovered from PPD and received training to deliver the intervention. The secondary objective of the RCT is to determine if the intervention can effectively treat its common comorbidities (anxiety) and complications (parenting stress, social support, mother-infant relationship, and infant temperament) and whether the intervention is cost-effective. 170 mothers/birthing parents will take part in the study with 50% being randomly assigned to the intervention group. All participants complete online questionnaires at 3 time points: baseline (T1), 9 weeks later (T2-immediately post-intervention in the experimental group to assess effectiveness) and 6 months later (T3-intervention durability).

ELIGIBILITY:
Inclusion Criteria:

Mothers or birthing parents, 18 years old, have an infant under 12 months of age at recruitment, fluent in written/spoken English, have a Edinburgh Postnatal Depression Scale (EPDS) score ≥10 and live in Ontario, Canada.

Exclusion Criteria:

Bipolar, psychotic, or current substance use disorders and borderline personality disorder as assessed during screening when study coordinator administers the Mini International Neuropsychiatric Interview (MINI).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum Depression | 9 weeks (post treatment/intervention)
  PPD is best conceptualized as a continuous construct with its impact operating across a continuum of severity. The primary outcome is change in PPD symptoms at 9 weeks (i.e., immediately post-treatment). This will be measured using the Edinburgh Postnatal Depression Scale (EPDS), a gold standard measure of PPD symptoms used commonly in research and clinical settings. The EPDS has 10 items scored on a scale 0-3. Scores range from 0-30, with higher scores indicating more severe depression symptoms. The EPDS will be examined as a continuous outcome. Changes in score of 4 or more points is considered clinically meaningful improvement.
Major Depressive Disorder | 9 weeks (post treatment/intervention)
  We will compare DSM-5-defined major depressive disorder (MDD) using the Mini International Neuropsychiatric Interview (MINI). This interview will be administered by telephone at T2-T3. Symptoms must be present every day or nearly every day for a period of at least 2 weeks and include at least one of: depressed mood most of the day, markedly diminished interest or pleasure in all or almost all activities. There must be a total of five symptoms including the previous two criteria and the following five criteria: significant unintentional weight change or appetite change; insomnia or hypersomnia; psychomotor agitation or retardation; fatigue; feelings of worthlessness or inappropriate or excessive guilt; decreased ability to concentrate or make decisions; recurrent thoughts of death or suicidal ideation.
Major Depressive Disorder | 6 months (durability of intervention effects)
  We will compare DSM-5-defined major depressive disorder (MDD) using the Mini International Neuropsychiatric Interview (MINI). This interview will be administered by telephone at T2-T3. Symptoms must be present every day or nearly every day for a period of at least 2 weeks and include at least one of: depressed mood most of the day, markedly diminished interest or pleasure in all or almost all activities. There must be a total of five symptoms including the previous two criteria and the following five criteria: significant unintentional weight change or appetite change; insomnia or hypersomnia; psychomotor agitation or retardation; fatigue; feelings of worthlessness or inappropriate or excessive guilt; decreased ability to concentrate or make decisions; recurrent thoughts of death or suicidal ideation.
Postpartum Depression | 6 months (durability of intervention effects)
  PPD is best conceptualized as a continuous construct with its impact operating across a continuum of severity. The primary outcome is change in PPD symptoms 6 months later (i.e., to assess durability of intervention effects). This will be measured using the Edinburgh Postnatal Depression Scale (EPDS), a gold standard measure of PPD symptoms used commonly in research and clinical settings. The EPDS has 10 items scored on a scale 0-3. Scores range from 0-30, with higher scores indicating more severe depression symptoms. The EPDS will be examined as a continuous outcome. Changes in score of 4 or more points is considered clinically meaningful improvement.

SECONDARY OUTCOMES:
Parenting Stress | 9 weeks (post treatment/intervention)
  The PSI-SF (Parenting Stress Index-Short Form ) is a 36-item self-scoring measure of parenting stress. It has 3 subscales: Parental distress, parent-child dysfunctional interaction and difficult child. Items are scored on a 5-point Likert scale. Higher scores indicate higher parental stress.
Parenting Stress | 6 months (durability of intervention effects)
  The PSI-SF (Parenting Stress Index-Short Form ) is a 36-item self-scoring measure of parenting stress. It has 3 subscales: Parental distress, parent-child dysfunctional interaction and difficult child. Items are scored on a 5-point Likert scale. Higher scores indicate higher parental stress.
Healthcare Resource Utilization Questionnaire | 9 weeks (post treatment/intervention)
  Healthcare resource utilization data will be collected using a questionnaire used in prior work and adapted for the postpartum period based on the Canadian Community Health Survey and Service Use and Resources Form. Participants will be asked to provide information on health care resource use including diagnosis and procedures, medications, hospital stays, physician and ER visits and the use of all other services (including those related to mental health). The investigators will measure resources consumed from the perspective of public health care payer and corresponding unit costs will be calculated using provincial billing rates.
Healthcare Resource Utilization Questionnaire | 6 months (durability of intervention effects)
  Healthcare resource utilization data will be collected using a questionnaire used in prior work and adapted for the postpartum period based on the Canadian Community Health Survey and Service Use and Resources Form. Participants will be asked to provide information on health care resource use including diagnosis and procedures, medications, hospital stays, physician and ER visits and the use of all other services (including those related to mental health). The investigators will measure resources consumed from the perspective of public health care payer and corresponding unit costs will be calculated using provincial billing rates.
Other Psychiatric Disorders | 9 weeks (post treatment/intervention)
  The Mini International Neuropsychiatric Interview (MINI) will be administered at T2 and T3 to provide information on the presence or absence of the major Axis 1 psychiatric disorders in the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM 5) at these time points. This will be administered by phone by a research assistant and will include the following modules: Major Depressive Episode; Major Depressive Disorder; Panic Disorder; Agoraphobia; Social Anxiety Disorder (Social Phobia); Obsessive-Compulsive Disorder; Posttraumatic Stress Disorder; Alcohol Use Disorder; Substance Use Disorder (Non-alcohol); Generalized Anxiety Disorder with extra screening questions for Psychosis.
Other Psychiatric Disorders | 6 months (durability of intervention effects)
  The Mini International Neuropsychiatric Interview (MINI) will be administered at T2 and T3 to provide information on the presence or absence of the major Axis 1 psychiatric disorders in the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM 5) at these time points. This will be administered by phone by a research assistant and will include the following modules: Major Depressive Episode; Major Depressive Disorder; Panic Disorder; Agoraphobia; Social Anxiety Disorder (Social Phobia); Obsessive-Compulsive Disorder; Posttraumatic Stress Disorder; Alcohol Use Disorder; Substance Use Disorder (Non-alcohol); Generalized Anxiety Disorder with extra screening questions for Psychosis.
Postpartum Anxiety | 9 weeks (post treatment/intervention)
  The GAD-7 (General Anxiety Disorder-7) is a reliable and valid 7-item self-report scale that assesses the symptoms of generalized anxiety disorder, the most common PPD comorbidity. Total score for the seven items ranges from 0-21 with a higher score indicating more severe anxiety symptoms.
Postpartum Anxiety | 6 months (durability of intervention effects)
  The GAD-7 (General Anxiety Disorder-7) is a reliable and valid 7-item self-report scale that assesses the symptoms of generalized anxiety disorder, the most common PPD comorbidity. Total score for the seven items ranges from 0-21 with a higher score indicating more severe anxiety symptoms.
Social Support | 9 weeks (post treatment/intervention)
  The MSPSS (Multidimensional Scale of Perceived Social Support) is a 12-item self-report scale designed to measure perceived social support from three sources: family, friends and partner. Each item is rated 1-7 with 1 very strongly disagree and 7 very strongly agree. Higher scores could be considered as having higher levels of support.
Social Support | 6 months (durability of intervention effects)
  The MSPSS (Multidimensional Scale of Perceived Social Support) is a 12-item self-report scale designed to measure perceived social support from three sources: family, friends and partner. Each item is rated 1-7 with 1 very strongly disagree and 7 very strongly agree. Higher scores could be considered as having higher levels of support.
Infant Temperament | 6 months (durability of intervention effects)
  The Infant Behavior Questionnaire - Revised (Very Short Form) is a parent report measure of infant temperament. The IBQ-R (Very Short Form) consists of 37 items answered on a 7-point scale (1-7) and assess 3 factors: Positive Affectivity/Surgency with 13 items, Negative Emotionality with 12 items and Orienting/Regulatory Capacity with 12 items. Higher scores indicate greater alignment with the domain.
Infant Temperament | 9 weeks (post treatment/intervention)
  The Infant Behavior Questionnaire - Revised (Very Short Form) is a parent report measure of infant temperament. The IBQ-R (Very Short Form) consists of 37 items answered on a 7-point scale (1-7) and assess 3 factors: Positive Affectivity/Surgency with 13 items, Negative Emotionality with 12 items and Orienting/Regulatory Capacity with 12 items. Higher scores indicate greater alignment with the domain.
Mother-Infant Relationship | 9 weeks (post treatment/intervention)
  The PBQ (Postpartum Bonding Questionnaire) is a 25-item maternal report measure that assesses four aspects of maternal-infant relations: (1) bonding, (2) rejection and anger towards the infant, (3) infant-focused anxiety and (4) incipient abuse. Subscales 1-3 will be explored as a continuous outcome using subscale total score. Respondents respond to each statement based on a 6-point scale, with total scale scores ranging from 0-125, with a higher cumulative score indicating more severe bonding disturbances. Each item is scored on a scale of 0-5 with higher scores suggestive of more problems. Mother-infant bonding will be measured as a continuous and dichotomous outcome, using cut-off scores for each subscale indicting bonding disorders. Cutoff values of 12 for the bonding subscale, 17 for rejection and anger, and 10 for infant-focused anxiety have been proposed to define bonding disorders in each category.
Mother-Infant Relationship | 6 months (durability of intervention effects)
  The PBQ (Postpartum Bonding Questionnaire) is a 25-item maternal report measure that assesses four aspects of maternal-infant relations: (1) bonding, (2) rejection and anger towards the infant, (3) infant-focused anxiety and (4) incipient abuse. Subscales 1-3 will be explored as a continuous outcome using subscale total score. Respondents respond to each statement based on a 6-point scale, with total scale scores ranging from 0-125, with a higher cumulative score indicating more severe bonding disturbances. Each item is scored on a scale of 0-5 with higher scores suggestive of more problems. Mother-infant bonding will be measured as a continuous and dichotomous outcome, using cut-off scores for each subscale indicting bonding disorders. Cutoff values of 12 for the bonding subscale, 17 for rejection and anger, and 10 for infant-focused anxiety have been proposed to define bonding disorders in each category.
Postpartum Anxiety | 9 weeks (post treatment/intervention)
  Postpartum Anxiety as a maternal comorbidity is a secondary outcome measure and the DSM-5 defined generalized anxiety disorder (GAD) will be compared using the Mini International Neuropsychiatric Interview (MINI). The GAD module will be part of the full MINI administered during screening and then administered again at T2 and T3 by phone by a research assistant. Excessive worry/anxiety about several routine things must be present most days in the preceding 6 months, anxiety/worry must be difficult to control as well as significantly disrupt social, work or relationship functions or cause significant distress. In order to meet the criteria for a Generalized Anxiety Disorder (current) to be present, three or more of the following must also be present in previous 6 months in addition to the previous three criteria: feel restless, keyed up or on edge; muscle tension; difficulties concentrating; irritability; sleep difficulties.
Postpartum Anxiety | 6 months (durability of intervention effects)
  Postpartum Anxiety as a maternal comorbidity is a secondary outcome measure and the DSM-5 defined generalized anxiety disorder (GAD) will be compared using the Mini International Neuropsychiatric Interview (MINI). The GAD module will be part of the full MINI administered during screening and then administered again at T2 and T3 by phone by a research assistant. Excessive worry/anxiety about several routine things must be present most days in the preceding 6 months, anxiety/worry must be difficult to control as well as significantly disrupt social, work or relationship functions or cause significant distress. In order to meet the criteria for a Generalized Anxiety Disorder (current) to be present, three or more of the following must also be present in previous 6 months in addition to the previous three criteria: feel restless, keyed up or on edge; muscle tension; difficulties concentrating; irritability; sleep difficulties.
EQ-5D-5L | 9-week (post treatment/intervention)
  A utility-based health-related quality of life self-report instrument consisting of five questions (scale of 1-5) covering mobility, self-care, usual activities, pain/discomfort and depression/anxiety. Lower scores indicate less problems. Quality of Life will be calculated using the Canadian scoring algorithm by multiplying the health utility for the corresponding time period (ie. area under the curve approach)
EQ-5D-5L | 6-month (durability of intervention effects)
  A utility-based health-related quality of life self-report instrument consisting of five questions (scale of 1-5) covering mobility, self-care, usual activities, pain/discomfort and depression/anxiety. Lower scores indicate less problems. Quality of Life will be calculated using the Canadian scoring algorithm by multiplying the health utility for the corresponding time period (ie. area under the curve approach)

OTHER OUTCOMES:
Fidelity of Intervention Delivery | Weekly during the 9-week intervention
  The fidelity with which the PHN/Peers deliver the 9-week CBT intervention will be assessed using measures of adherence and competence that were developed for evaluating delivery of the 9-week CBT groups. Each of the weekly CBT groups will be digitally recorded and trained raters will rate the adherence to the intervention model and competence with which the PHN/Peers deliver the intervention.
Assess Participant Satisfaction | 9-week (post treatment/intervention)
  The Client Satisfaction Questionnaire-8 (CSQ-8) is an 8-item measure that measures and assesses consumer satisfaction with health and human services. Items are scored on a 4-point scale and total scores range from 8-32, with higher scores indicating greater satisfaction. This will only be completed by participants who complete the 9-week CBT group, immediately after they participate in the intervention.
Psychotherapy Experience | 9 weeks (post treatment/intervention)
  Study participants will complete this questionnaire at T2 (past 9 weeks) and T3 (past 6 months) answering questions if they received any type of talking therapy or psychotherapy (ie. Cognitive Behavioural Therapy, Group Therapy) other than the group CBT sessions they may have attended as part of the research study. The questions ask about type of therapy received, why it was received, the number of sessions received and the date started and stopped. This information will be used as part of the sub-group analysis to examine the impact of other therapies on the intervention effectiveness.
Psychotherapy Experience | 6 months (durability of intervention effects)
  Study participants will complete this questionnaire at T2 (past 9 weeks) and T3 (past 6 months) answering questions if they received any type of talking therapy or psychotherapy (ie. Cognitive Behavioural Therapy, Group Therapy) other than the group CBT sessions they may have attended as part of the research study. The questions ask about type of therapy received, why it was received, the number of sessions received and the date started and stopped. This information will be used as part of the sub-group analysis to examine the impact of other therapies on the intervention effectiveness.
Personal Attributes | 9 weeks (post treatment/intervention)
  A 24-item self-report measure of gender identity. We will examine the moderating effect of its instrumentality and expressivity scales, as well as self-identified gender identity on our outcomes
Personal Attributes | 6 months (durability of intervention effects)
  A 24-item self-report measure of gender identity. We will examine the moderating effect of its instrumentality and expressivity scales, as well as self-identified gender identity on our outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Van Lieshout, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to other researchers

REFERENCES:
- [Background] Gavin NI, Gaynes BN, Lohr KN, Meltzer-Brody S, Gartlehner G, Swinson T. Perinatal depression: a systematic review of prevalence and incidence. Obstet Gynecol. 2005 Nov;106(5 Pt 1):1071-83. doi: 10.1097/01.AOG.0000183597.31630.db. PMID 16260528
- [Background] Lanes A, Kuk JL, Tamim H. Prevalence and characteristics of postpartum depression symptomatology among Canadian women: a cross-sectional study. BMC Public Health. 2011 May 11;11:302. doi: 10.1186/1471-2458-11-302. PMID 21569372
- [Background] Zanardo V, Manghina V, Giliberti L, Vettore M, Severino L, Straface G. Psychological impact of COVID-19 quarantine measures in northeastern Italy on mothers in the immediate postpartum period. Int J Gynaecol Obstet. 2020 Aug;150(2):184-188. doi: 10.1002/ijgo.13249. Epub 2020 Jun 16. PMID 32474910
- [Background] Lakshmin P. Experts Fear Increase in Postpartum Mood and Anxiety Disorders. The New York Times [Internet]. 2020 https://wwwnytimes.com/2020/05/27/parenting/coronavirus-postpartum-depressionanxiety.html?smid=tw-share
- [Background] Goodman SH, Rouse MH, Connell AM, Broth MR, Hall CM, Heyward D. Maternal depression and child psychopathology: a meta-analytic review. Clin Child Fam Psychol Rev. 2011 Mar;14(1):1-27. doi: 10.1007/s10567-010-0080-1. PMID 21052833
- [Background] Lovejoy MC, Graczyk PA, O'Hare E, Neuman G. Maternal depression and parenting behavior: a meta-analytic review. Clin Psychol Rev. 2000 Aug;20(5):561-92. doi: 10.1016/s0272-7358(98)00100-7. PMID 10860167
- [Background] Barry TJ, Murray L, Fearon RM, Moutsiana C, Cooper P, Goodyer IM, Herbert J, Halligan SL. Maternal postnatal depression predicts altered offspring biological stress reactivity in adulthood. Psychoneuroendocrinology. 2015 Feb;52:251-60. doi: 10.1016/j.psyneuen.2014.12.003. Epub 2014 Dec 9. PMID 25544737
- [Background] Murray L, Fearon P, Cooper P. Postnatal Depression, Mother-Infant Interactions, and Child Development. Identifying Perinatal Depression and Anxiety. John Wiley & Sons, Ltd; 2015:139-164. doi:10.1002/9781118509722.ch9
- [Background] Burke L. The impact of maternal depression on familial relationships. Int Rev Psychiatry. 2003 Aug;15(3):243-55. doi: 10.1080/0954026031000136866. PMID 15276963
- [Background] Grace SL, Evindar A, Stewart DE. The effect of postpartum depression on child cognitive development and behavior: a review and critical analysis of the literature. Arch Womens Ment Health. 2003 Nov;6(4):263-74. doi: 10.1007/s00737-003-0024-6. PMID 14628179
- [Background] Halligan SL, Murray L, Martins C, Cooper PJ. Maternal depression and psychiatric outcomes in adolescent offspring: a 13-year longitudinal study. J Affect Disord. 2007 Jan;97(1-3):145-54. doi: 10.1016/j.jad.2006.06.010. Epub 2006 Jul 24. PMID 16863660
- [Background] O'Hara MW, McCabe JE. Postpartum depression: current status and future directions. Annu Rev Clin Psychol. 2013;9:379-407. doi: 10.1146/annurev-clinpsy-050212-185612. Epub 2013 Feb 1. PMID 23394227
- [Background] Bauer A, Knapp M, Adelaja B. Best practice for perinatal mental health care: the economic case. PSSRU Rep. 2016.
- [Background] Krzeczkowski JE, Schmidt LA, Van Lieshout RJ. Changes in infant emotion regulation following maternal cognitive behavioral therapy for postpartum depression. Depress Anxiety. 2021 Apr;38(4):412-421. doi: 10.1002/da.23130. Epub 2021 Jan 19. PMID 33464686
- [Background] Letourneau NL, Dennis CL, Cosic N, Linder J. The effect of perinatal depression treatment for mothers on parenting and child development: A systematic review. Depress Anxiety. 2017 Oct;34(10):928-966. doi: 10.1002/da.22687. Epub 2017 Sep 29. PMID 28962068
- [Background] Van Lieshout RJ, Layton H, Savoy CD, Brown JSL, Ferro MA, Streiner DL, Bieling PJ, Feller A, Hanna S. Effect of Online 1-Day Cognitive Behavioral Therapy-Based Workshops Plus Usual Care vs Usual Care Alone for Postpartum Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Nov 1;78(11):1200-1207. doi: 10.1001/jamapsychiatry.2021.2488. PMID 34495285
- [Background] MacQueen GM, Frey BN, Ismail Z, Jaworska N, Steiner M, Lieshout RJ, Kennedy SH, Lam RW, Milev RV, Parikh SV, Ravindran AV; CANMAT Depression Work Group. Canadian Network for Mood and Anxiety Treatments (CANMAT) 2016 Clinical Guidelines for the Management of Adults with Major Depressive Disorder: Section 6. Special Populations: Youth, Women, and the Elderly. Can J Psychiatry. 2016 Sep;61(9):588-603. doi: 10.1177/0706743716659276. Epub 2016 Aug 2. PMID 27486149
- [Background] Surveillance report 2017 - Antenatal and postnatal mental health: clinical management and service guidance (2014) NICE guideline CG192 [Internet]. London: National Institute for Health and Care Excellence (NICE); 2017 Jun 8. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK550943/ PMID 31841290
- [Background] Siu AL; US Preventive Services Task Force (USPSTF); Bibbins-Domingo K, Grossman DC, Baumann LC, Davidson KW, Ebell M, Garcia FA, Gillman M, Herzstein J, Kemper AR, Krist AH, Kurth AE, Owens DK, Phillips WR, Phipps MG, Pignone MP. Screening for Depression in Adults: US Preventive Services Task Force Recommendation Statement. JAMA. 2016 Jan 26;315(4):380-7. doi: 10.1001/jama.2015.18392. PMID 26813211
- [Background] Elkhodr S, Saba M, O'Reilly C, Saini B. The role of community pharmacists in the identification and ongoing management of women at risk for perinatal depression: A qualitative study. Int J Soc Psychiatry. 2018 Feb;64(1):37-48. doi: 10.1177/0020764017746198. Epub 2017 Dec 8. PMID 29219031
- [Background] National Institute for Health and Care Excellence. Common Mental Health Disorders: Identification and Pathways to Care. NICE clinical guideline CG123. London: NICE; 2011. Available from: https://www.nice.org.uk/guidance/cg123
- [Background] Hadfield H, Wittkowski A. Women's Experiences of Seeking and Receiving Psychological and Psychosocial Interventions for Postpartum Depression: A Systematic Review and Thematic Synthesis of the Qualitative Literature. J Midwifery Womens Health. 2017 Nov;62(6):723-736. doi: 10.1111/jmwh.12669. Epub 2017 Dec 6. PMID 29210501
- [Background] Trevillion K, Ryan EG, Pickles A, Heslin M, Byford S, Nath S, Bick D, Milgrom J, Mycroft R, Domoney J, Pariante C, Hunter MS, Howard LM. An exploratory parallel-group randomised controlled trial of antenatal Guided Self-Help (plus usual care) versus usual care alone for pregnant women with depression: DAWN trial. J Affect Disord. 2020 Jan 15;261:187-197. doi: 10.1016/j.jad.2019.10.013. Epub 2019 Oct 12. PMID 31634678
- [Background] Tsai Z, Kiss A, Nadeem S, Sidhom K, Owais S, Faltyn M, Lieshout RJV. Evaluating the effectiveness and quality of mobile applications for perinatal depression and anxiety: A systematic review and meta-analysis. J Affect Disord. 2022 Jan 1;296:443-453. doi: 10.1016/j.jad.2021.09.106. Epub 2021 Oct 6. PMID 34624434
- [Background] Singla DR, Ratjen C, Krishna RN, Fuhr DC, Patel V. Peer supervision for assuring the quality of non-specialist provider delivered psychological intervention: Lessons from a trial for perinatal depression in Goa, India. Behav Res Ther. 2020 Jul;130:103533. doi: 10.1016/j.brat.2019.103533. Epub 2019 Dec 17. PMID 31870496
- [Background] Dennis CL, Chung-Lee L. Postpartum depression help-seeking barriers and maternal treatment preferences: a qualitative systematic review. Birth. 2006 Dec;33(4):323-31. doi: 10.1111/j.1523-536X.2006.00130.x. PMID 17150072
- [Background] Bryan AE, Arkowitz H. Meta-analysis of the effects of peer-administered psychosocial interventions on symptoms of depression. Am J Community Psychol. 2015 Jun;55(3-4):455-71. doi: 10.1007/s10464-015-9718-y. PMID 25861883
- [Background] Goodman JH. Women's attitudes, preferences, and perceived barriers to treatment for perinatal depression. Birth. 2009 Mar;36(1):60-9. doi: 10.1111/j.1523-536X.2008.00296.x. PMID 19278385
- [Background] Newman TC, Hirst J, Darwin Z. What enables or prevents women with depressive symptoms seeking help in the postnatal period? Br J Midwifery. 2019;27(4):219-227. doi:10.12968/bjom.2019.27.4.219
- [Background] Bickman L. Practice Makes Perfect and Other Myths about Mental Health Services. Am Psychol. 1999;54(11):965-978. doi:10.1037/h0088206
- [Background] Dennis CL, Falah-Hassani K, Shiri R. Prevalence of antenatal and postnatal anxiety: systematic review and meta-analysis. Br J Psychiatry. 2017 May;210(5):315-323. doi: 10.1192/bjp.bp.116.187179. Epub 2017 Mar 16. PMID 28302701
- [Background] Montgomery EC, Kunik ME, Wilson N, Stanley MA, Weiss B. Can paraprofessionals deliver cognitive-behavioral therapy to treat anxiety and depressive symptoms? Bull Menninger Clin. 2010 Winter;74(1):45-62. doi: 10.1521/bumc.2010.74.1.45. PMID 20235623
- [Background] Holopainen D. The experience of seeking help for postnatal depression. Aust J Adv Nurs. 2002 Mar-May;19(3):39-44. PMID 12002628
- [Background] Prevatt BS, Lowder EM, Desmarais SL. Peer-support intervention for postpartum depression: Participant satisfaction and program effectiveness. Midwifery. 2018 Sep;64:38-47. doi: 10.1016/j.midw.2018.05.009. Epub 2018 May 31. PMID 29908406
- [Background] Montgomery P, Mossey S, Adams S, Bailey PH. Stories of women involved in a postpartum depression peer support group. Int J Ment Health Nurs. 2012 Dec;21(6):524-32. doi: 10.1111/j.1447-0349.2012.00828.x. Epub 2012 Jun 27. PMID 22738350
- [Background] Mead S, Hilton D, Curtis L. Peer support: a theoretical perspective. Psychiatr Rehabil J. 2001 Fall;25(2):134-41. doi: 10.1037/h0095032. PMID 11769979
- [Background] Solomon P. Peer support/peer provided services underlying processes, benefits, and critical ingredients. Psychiatr Rehabil J. 2004 Spring;27(4):392-401. doi: 10.2975/27.2004.392.401. PMID 15222150
- [Background] Resnick SG, Rosenheck RA. Integrating peer-provided services: a quasi-experimental study of recovery orientation, confidence, and empowerment. Psychiatr Serv. 2008 Nov;59(11):1307-14. doi: 10.1176/ps.2008.59.11.1307. PMID 18971407
- [Background] Letourneau N, Duffett-Leger L, Stewart M, Hegadoren K, Dennis CL, Rinaldi CM, Stoppard J. Canadian mothers' perceived support needs during postpartum depression. J Obstet Gynecol Neonatal Nurs. 2007 Sep-Oct;36(5):441-9. doi: 10.1111/j.1552-6909.2007.00174.x. PMID 17880314
- [Background] Singla DR, Lemberg-Pelly S, Lawson A, Zahedi N, Thomas-Jacques T, Dennis CL. Implementing Psychological Interventions Through Nonspecialist Providers and Telemedicine in High-Income Countries: Qualitative Study from a Multistakeholder Perspective. JMIR Ment Health. 2020 Aug 27;7(8):e19271. doi: 10.2196/19271. PMID 32852281
- [Background] Noonan M, Galvin R, Doody O, Jomeen J. A qualitative meta-synthesis: public health nurses role in the identification and management of perinatal mental health problems. J Adv Nurs. 2017 Mar;73(3):545-557. doi: 10.1111/jan.13155. Epub 2016 Oct 20. PMID 27653522
- [Background] Layton H, Bendo D, Amani B, Bieling PJ, Van Lieshout RJ. Public health nurses' experiences learning and delivering a group cognitive behavioral therapy intervention for postpartum depression. Public Health Nurs. 2020 Nov;37(6):863-870. doi: 10.1111/phn.12807. Epub 2020 Sep 13. PMID 32924183
- [Background] Healthy Human Development Table. Perinatal Mental Health Toolkit for Ontario Public Health Units. 2018.
- [Background] Austin M, Highet N and the EWG. Mental Health Care in the Perinatal Period: Australian Clinical Practice Guideline. 2017:1-121.
- [Background] Nillni YI, Mehralizade A, Mayer L, Milanovic S. Treatment of depression, anxiety, and trauma-related disorders during the perinatal period: A systematic review. Clin Psychol Rev. 2018 Dec;66:136-148. doi: 10.1016/j.cpr.2018.06.004. Epub 2018 Jun 9. PMID 29935979
- [Background] Cuijpers P, Van Straten A, Warmerdam L. Are individual and group treatments equally effective in the treatment of depression in adults? A meta-analysis. Eur J Psychiatry. 2008;22(1):38-51. doi:10.4321/S0213-61632008000100005
- [Background] Sockol LE. A systematic review of the efficacy of cognitive behavioral therapy for treating and preventing perinatal depression. J Affect Disord. 2015 May 15;177:7-21. doi: 10.1016/j.jad.2015.01.052. Epub 2015 Feb 2. PMID 25743368
- [Background] Butler AC, Chapman JE, Forman EM, Beck AT. The empirical status of cognitive-behavioral therapy: a review of meta-analyses. Clin Psychol Rev. 2006 Jan;26(1):17-31. doi: 10.1016/j.cpr.2005.07.003. Epub 2005 Sep 30. PMID 16199119
- [Background] Singla DR, Lawson A, Kohrt BA, Jung JW, Meng Z, Ratjen C, Zahedi N, Dennis CL, Patel V. Implementation and Effectiveness of Nonspecialist-Delivered Interventions for Perinatal Mental Health in High-Income Countries: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2021 May 1;78(5):498-509. doi: 10.1001/jamapsychiatry.2020.4556. PMID 33533904
- [Background] Honey KL, Bennett P, Morgan M. A brief psycho-educational group intervention for postnatal depression. Br J Clin Psychol. 2002 Nov;41(Pt 4):405-9. doi: 10.1348/014466502760387515. PMID 12437794
- [Background] Van Lieshout RJ, Layton H, Savoy CD, Haber E, Feller A, Biscaro A, Bieling PJ, Ferro MA. Public Health Nurse-delivered Group Cognitive Behavioural Therapy for Postpartum Depression: A Randomized Controlled Trial. Can J Psychiatry. 2022 Jun;67(6):432-440. doi: 10.1177/07067437221074426. Epub 2022 Jan 21. PMID 35060398
- [Background] Huh K, Layton H, Savoy CD, Ferro MA, Bieling PJ, Hicks A, Van Lieshout RJ. Online Public Health Nurse-Delivered Group Cognitive Behavioral Therapy for Postpartum Depression: A Randomized Controlled Trial During the COVID-19 Pandemic. J Clin Psychiatry. 2023 Jul 24;84(5):22m14726. doi: 10.4088/JCP.22m14726. PMID 37498661
- [Background] Dennis CL. The effect of peer support on postpartum depression: a pilot randomized controlled trial. Can J Psychiatry. 2003 Mar;48(2):115-24. doi: 10.1177/070674370304800209. PMID 12655910
- [Background] Dennis CL, Hodnett E, Kenton L, Weston J, Zupancic J, Stewart DE, Kiss A. Effect of peer support on prevention of postnatal depression among high risk women: multisite randomised controlled trial. BMJ. 2009 Jan 15;338:a3064. doi: 10.1136/bmj.a3064. PMID 19147637
- [Background] Letourneau N, Stewart M, Dennis CL, Hegadoren K, Duffett-Leger L, Watson B. Effect of home-based peer support on maternal-infant interactions among women with postpartum depression: a randomized, controlled trial. Int J Ment Health Nurs. 2011 Oct;20(5):345-57. doi: 10.1111/j.1447-0349.2010.00736.x. Epub 2011 Mar 8. PMID 21385294
- [Background] Gjerdingen DK, McGovern P, Pratt R, Johnson L, Crow S. Postpartum doula and peer telephone support for postpartum depression: a pilot randomized controlled trial. J Prim Care Community Health. 2013 Jan;4(1):36-43. doi: 10.1177/2150131912451598. Epub 2012 Jun 20. PMID 23799688
- [Background] Shorey S, Chee CYI, Ng ED, Lau Y, Dennis CL, Chan YH. Evaluation of a Technology-Based Peer-Support Intervention Program for Preventing Postnatal Depression (Part 1): Randomized Controlled Trial. J Med Internet Res. 2019 Aug 29;21(8):e12410. doi: 10.2196/12410. PMID 31469084
- [Background] Fuhr DC, Weobong B, Lazarus A, Vanobberghen F, Weiss HA, Singla DR, Tabana H, Afonso E, De Sa A, D'Souza E, Joshi A, Korgaonkar P, Krishna R, Price LN, Rahman A, Patel V. Delivering the Thinking Healthy Programme for perinatal depression through peers: an individually randomised controlled trial in India. Lancet Psychiatry. 2019 Feb;6(2):115-127. doi: 10.1016/S2215-0366(18)30466-8. PMID 30686385
- [Background] Sikander S, Ahmad I, Atif N, Zaidi A, Vanobberghen F, Weiss HA, Nisar A, Tabana H, Ain QU, Bibi A, Bilal S, Bibi T, Liaqat R, Sharif M, Zulfiqar S, Fuhr DC, Price LN, Patel V, Rahman A. Delivering the Thinking Healthy Programme for perinatal depression through volunteer peers: a cluster randomised controlled trial in Pakistan. Lancet Psychiatry. 2019 Feb;6(2):128-139. doi: 10.1016/S2215-0366(18)30467-X. PMID 30686386
- [Background] Amani B, Merza D, Savoy C, Streiner D, Bieling P, Ferro MA, Van Lieshout RJ. Peer-Delivered Cognitive-Behavioral Therapy for Postpartum Depression: A Randomized Controlled Trial. J Clin Psychiatry. 2021 Nov 9;83(1):21m13928. doi: 10.4088/JCP.21m13928. PMID 34758210
- [Background] Merza D, Amani B, Savoy C, Babiy Z, Bieling PJ, Streiner DL, Ferro MA, Van Lieshout RJ. Online peer-delivered group cognitive-behavioral therapy for postpartum depression: A randomized controlled trial. Acta Psychiatr Scand. 2024 Nov;150(5):422-432. doi: 10.1111/acps.13611. Epub 2023 Aug 31. PMID 37649448
- [Background] Merza D, Layton H, Savoy C, Babiy Z, Campbell M, Bieling PJ, Brown JSL, Van Lieshout RJ. Online Peer-Delivered 1-Day Cognitive Behavioral Therapy-Based Workshops for Postpartum Depression: A Pilot Study. J Clin Psychiatry. 2023 Jan 2;84(1):22br14574. doi: 10.4088/JCP.22br14574. No abstract available. PMID 36602928
- [Background] Taylor D. Effectiveness of professional--peer group treatment: symptom management for women with PMS. Res Nurs Health. 1999 Dec;22(6):496-511. doi: 10.1002/(sici)1098-240x(199912)22:63.0.co;2-2. PMID 10625865
- [Background] Goldberg RW, Dickerson F, Lucksted A, Brown CH, Weber E, Tenhula WN, Kreyenbuhl J, Dixon LB. Living well: an intervention to improve self-management of medical illness for individuals with serious mental illness. Psychiatr Serv. 2013 Jan;64(1):51-7. doi: 10.1176/appi.ps.201200034. PMID 23070062
- [Background] Muralidharan A, Brown CH, E Peer J, A Klingaman E, M Hack S, Li L, Walsh MB, Goldberg RW. Living Well: An Intervention to Improve Medical Illness Self-Management Among Individuals With Serious Mental Illness. Psychiatr Serv. 2019 Jan 1;70(1):19-25. doi: 10.1176/appi.ps.201800162. Epub 2018 Oct 24. PMID 30353790
- [Background] Chibanda D, Shetty AK, Tshimanga M, Woelk G, Stranix-Chibanda L, Rusakaniko S. Group problem-solving therapy for postnatal depression among HIV-positive and HIV-negative mothers in Zimbabwe. J Int Assoc Provid AIDS Care. 2014 Jul-Aug;13(4):335-41. doi: 10.1177/2325957413495564. PMID 23881909
- [Background] Cameron EE, Joyce KM, Delaquis CP, Reynolds K, Protudjer JLP, Roos LE. Maternal psychological distress & mental health service use during the COVID-19 pandemic. J Affect Disord. 2020 Nov 1;276:765-774. doi: 10.1016/j.jad.2020.07.081. Epub 2020 Jul 20. PMID 32736186
- [Background] Bartram M, Chodos H. Changing Directions, Changing Lives: The Mental Health Strategy for Canada. Can J Commun Ment Health. 2013;32:1-8. doi:10.7870/cjcmh-2013-001
- [Background] Van Lieshout RJ, Yang L, Haber E, Ferro MA. Evaluating the effectiveness of a brief group cognitive behavioural therapy intervention for perinatal depression. Arch Womens Ment Health. 2017 Feb;20(1):225-228. doi: 10.1007/s00737-016-0666-9. Epub 2016 Sep 10. PMID 27613531
- [Background] Van Lieshout RJ, Layton H, Feller A, Ferro MA, Biscaro A, Bieling PJ. Public health nurse delivered group cognitive behavioral therapy (CBT) for postpartum depression: A pilot study. Public Health Nurs. 2020 Jan;37(1):50-55. doi: 10.1111/phn.12664. Epub 2019 Sep 15. PMID 31523851
- [Background] Van Lieshout RJ, Layton H, Rangan M, Ferro MA, Brown JSL, Bieling PJ. Treating Postpartum Depression With 1-Day Cognitive Behavioural Therapy-Based Workshops. J Obstet Gynaecol Can. 2019 May;41(5):591-592. doi: 10.1016/j.jogc.2019.02.018. Epub 2019 Mar 9. No abstract available. PMID 30862440
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Beck AT, Steer RA, Brown G. Beck Depression Inventory-II. Psychological assessment. 1996.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] R Core Team. R: A Language and Environment for Statistical Computing [Internet]. Vienna, Austria; 2016. Available from: https://www.R-project.org/
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Ebert JF, Huibers L, Christensen B, Christensen MB. Paper- or Web-Based Questionnaire Invitations as a Method for Data Collection: Cross-Sectional Comparative Study of Differences in Response Rate, Completeness of Data, and Financial Cost. J Med Internet Res. 2018 Jan 23;20(1):e24. doi: 10.2196/jmir.8353. PMID 29362206
- [Background] Dillman, D.A., Smyth, J.D. CL. Internet, Phone, Maiol, and Mixed-Mode Surveys: The Tailored Design Method. 4th ed. Hoboken, NJ: Wiley; 2014.
- [Background] Meaney MJ. Perinatal Maternal Depressive Symptoms as an Issue for Population Health. Am J Psychiatry. 2018 Nov 1;175(11):1084-1093. doi: 10.1176/appi.ajp.2018.17091031. Epub 2018 Aug 2. PMID 30068258
- [Background] Sockol LE. A systematic review and meta-analysis of interpersonal psychotherapy for perinatal women. J Affect Disord. 2018 May;232:316-328. doi: 10.1016/j.jad.2018.01.018. Epub 2018 Feb 1. PMID 29501991
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Loyd BH, Abidin RR. Revision of the Parenting Stress Index. J Pediatr Psychol. 1985 Jun;10(2):169-77. doi: 10.1093/jpepsy/10.2.169. No abstract available. PMID 4020601
- [Background] Brockington IF, Fraser C, Wilson D. The Postpartum Bonding Questionnaire: a validation. Arch Womens Ment Health. 2006 Sep;9(5):233-42. doi: 10.1007/s00737-006-0132-1. Epub 2006 May 4. PMID 16673041
- [Background] Brockington IF, Oates J, George S, Turner D, Vostanis P, Sullivan M, et al. A screening questionnaire for mother-infant bonding disorders. Arch Womens Ment Health. 2001;3(4):133- 140.
- [Background] Zimet GD, Dahlem NW, Zimet SG, et al. The multidimensional scale of perceived social support. J Pers Assess. 1988;52(1):30-41. doi:10.1207/s15327752jpa5201_2
- [Background] Putnam SP, Helbig AL, Gartstein MA, Rothbart MK, Leerkes E. Development and assessment of short and very short forms of the infant behavior questionnaire-revised. J Pers Assess. 2014;96(4):445-58. doi: 10.1080/00223891.2013.841171. Epub 2013 Nov 9. PMID 24206185
- [Background] Helmreich RL, Spence JT, Wilhelm JA. A psychometric analysis of the Personal Attributes Questionnaire. Sex Roles. 1981;7:1097-1108. doi:10.1007/BF00287587
- [Background] Canadian Community Health Survey (CCHS). Questionnaire for Cycle 1.1. 2001.
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Crick K, Al Sayah F, Ohinmaa A, Johnson JA. Responsiveness of the anxiety/depression dimension of the 3- and 5-level versions of the EQ-5D in assessing mental health. Qual Life Res. 2018 Jun;27(6):1625-1633. doi: 10.1007/s11136-018-1828-1. Epub 2018 Mar 7. PMID 29516342
- [Background] Xie F, Pullenayegum E, Gaebel K, Bansback N, Bryan S, Ohinmaa A, Poissant L, Johnson JA; Canadian EQ-5D-5L Valuation Study Group. A Time Trade-off-derived Value Set of the EQ-5D-5L for Canada. Med Care. 2016 Jan;54(1):98-105. doi: 10.1097/MLR.0000000000000447. PMID 26492214
- [Background] Cliffe T, Beinart H, Cooper M. Development and Validation of a Short Version of the Supervisory Relationship Questionnaire. Clin Psychol Psychother. 2016 Jan-Feb;23(1):77-86. doi: 10.1002/cpp.1935. Epub 2014 Dec 11. PMID 25504780
- [Background] Milne DL, Reiser RP. SAGE. In: The Wiley International Handbook of Clinical Supervision. John Wiley & Sons, Ltd; 2014:402-415. doi:10.1002/9781118846360.ch18
- [Background] Hepner KA, Howard S, Paddock SM, Hunter SB, Osilla KC, Watkins KE. A Fidelity Coding Guide for a Group Cognitive Behavioral Therapy for Depression. RAND Corporation; 2011. https://www.rand.org/pubs/technical_reports/TR980.html
- [Background] Babiy Z, Merza D, Layton H, Bieling PJ, Van Lieshout RJ. Fidelity Assessment of Peer-Delivered Cognitive-Behavioral Therapy for Postpartum Depression. Am J Psychother. 2023 Dec 11;76(4):159-162. doi: 10.1176/appi.psychotherapy.20220060. Epub 2023 Aug 23. PMID 37608754
- [Background] McGuire-Snieckus R, McCabe R, Catty J, Hansson L, Priebe S. A new scale to assess the therapeutic relationship in community mental health care: STAR. Psychol Med. 2007 Jan;37(1):85-95. doi: 10.1017/S0033291706009299. Epub 2006 Nov 9. PMID 17094819
- [Background] Williams MT, Tellawi G, Wetterneck CT, Chapman LK. Recruitment of ethnoracial minorities for mental health research. Behav Ther. 2013;36(6):151-156.
- [Background] Waheed W, Hughes-Morley A, Woodham A, Allen G, Bower P. Overcoming barriers to recruiting ethnic minorities to mental health research: a typology of recruitment strategies. BMC Psychiatry. 2015 May 2;15:101. doi: 10.1186/s12888-015-0484-z. PMID 25934297
- [Background] Renert H, Russell-Mayhew S, Arthur N. Recruiting ethnically diverse participants into qualitative health research: Lessons learned. Qual Rep. 2013;18(12):1-13.
- [Background] Singer J, Willett J. Applied Longitudinal Data Analysis. Modeling Change and Event Occurrence. New York: Oxford University Press; 2003.
- [Background] Stekhoven DJ, Buhlmann P. MissForest--non-parametric missing value imputation for mixed-type data. Bioinformatics. 2012 Jan 1;28(1):112-8. doi: 10.1093/bioinformatics/btr597. Epub 2011 Oct 28. PMID 22039212
- [Background] Husereau D, Drummond M, Petrou S, Carswell C, Moher D, Greenberg D, Augustovski F, Briggs AH, Mauskopf J, Loder E; CHEERS Task Force. Consolidated Health Economic Evaluation Reporting Standards (CHEERS) statement. Int J Technol Assess Health Care. 2013 Apr;29(2):117-22. doi: 10.1017/S0266462313000160. Epub 2013 Apr 15. PMID 23587340
- [Background] Petrou S, Gray A. Economic evaluation alongside randomised controlled trials: design, conduct, analysis, and reporting. BMJ. 2011 Apr 7;342:d1548. doi: 10.1136/bmj.d1548. PMID 21474510
- [Background] Sandelowski M. Whatever happened to qualitative description? Res Nurs Health. 2000 Aug;23(4):334-40. doi: 10.1002/1098-240x(200008)23:43.0.co;2-g. PMID 10940958
- [Background] Palinkas LA, Horwitz SM, Green CA, Wisdom JP, Duan N, Hoagwood K. Purposeful Sampling for Qualitative Data Collection and Analysis in Mixed Method Implementation Research. Adm Policy Ment Health. 2015 Sep;42(5):533-44. doi: 10.1007/s10488-013-0528-y. PMID 24193818
- [Background] Dedoose Version 9.0.17. Cloud application for managing, analyzing, and presenting qualitative and mixed method research data (2021). Los Angeles, CA: SocioCultural Research Consultants, LLC www.dedoose.com
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937